CLINICAL TRIAL: NCT04610307
Title: EFFECT OF BUFFERED LOCAL ANESTHESIA ON PAIN DURING ARTERIOVEONUS FISTULA
Brief Title: EFFECT OF BUFFERED LOCAL ANESTHESIA ON PAIN IN ARETERIOVENOUS FISTULA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Combined Military Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Dr Anum Arif, Dr Anum Arif, Combined Military Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CMHLahore
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Pain, Procedural; Pain, Postoperative; Satisfaction, Patient
MeSH Terms: conditions — Pain, Procedural; Pain, Postoperative; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): patients receiving 1 % plain xylocaine
  Interventions: Procedure: buffered anesthesia
- intervention group (Experimental): patients receiving buffered 1 % xylocaine
  Interventions: Procedure: buffered anesthesia

INTERVENTIONS:
Procedure: buffered anesthesia — patients will undergo surgery under buffered local anesthesia

SUMMARY:
Pain and satisfaction score will be assessed at the end of surgery and compared in either of two groups

DETAILED DESCRIPTION:
All patients meeting inclusion criteria will be randomly enrolled in two groups. Intervention group will receive buffered lignocaine . at the end of procedure data will be recorded regarding pain VASscore and satisfaction score

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III
* Brachiocephalic arteriovenous fistula
* Radiocephalic arteriovenous fistula

Exclusion Criteria:

* basiic vein transposition
* redo surgery emergency surgery
* failure to understand the questionnnare

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
pain score | 60 minutes
  pain score on visual analog score on a scale of 0 to 10. 0 means no pain. 1 is least pain and 10 is maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- Combined Military Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No